CLINICAL TRIAL: NCT06410820
Title: Comparison of Ultrasound and Anatomical Landmark Method in Spinal Anesthesia for Elective Cesarean Section in Super Obese Parturients With BMI ≥ 50 kg/m2. A Randomized Controlled Trial
Brief Title: Ultrasound Guided Versus Land-mark Method for Spinal Anesthesia in Super Obesity Parturients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karaman Training and Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11-2022/03
Record Dates: First submitted 2024-04-04; First posted 2024-05-13 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-04

CONDITIONS: Obesity, Morbid
Keywords: Spinal Anesthesia; Cesarean Delivery; Ultrasound
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Allocation: Randomized Intervention Model: Parallel Assignment
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound method group (Active Comparator): The ultrasound-assisted technique will be used for spinal anesthesia performance.
  Interventions: Device: Procedure/Surgery: Ultrasound method group
- Landmark method group (Experimental): Land-mark assisted technique will be used for spinal anesthesia performance.
  Interventions: Device: Landmark method group

INTERVENTIONS:
Device: Procedure/Surgery: Ultrasound method group — In the operating room, all of the patients will receive standard monitoring. Scans will be made in logiditunal parasagittal and transverse midline views with ultrasound. Needle entry sites in the L2-L3 and L3-L4 intervals will be determined as the intersection of the longiditunal and transverse lines.
  When the spinal puncture operator is outside the room, Needle entry sites were marked for both groups.After skin marking, the pregnant woman will be asked to remain still and a subarachnoid puncture will be performed immediately. Spinal anesthesia will be administered with injection of intrathecal bupivacaine.
  Arms: Ultrasound method group
Device: Landmark method group — In the Landmark group, the injection site will be determined using the traditional method of palpating the posterior superior iliac spine.When the spinal puncture operator is outside the room, Needle entry sites were marked for both groups.After skin marking, the pregnant woman will be asked to remain still and a subarachnoid puncture will be performed immediately. Spinal anesthesia will be administered with injection of intrathecal bupivacaine.
  Arms: Landmark method group

SUMMARY:
This study will investigate whether an ultrasound-assisted technique is better than a classical land-mark technique to facilitate spinal anesthesia in the sitting position in super obese pregnant women with BMI ≥ 50 who will undergo elective cesarean section.

The primary objective of this study is the rate of successful dural puncture at the first attempt. It was assumed that ultrasound could facilitate neuraxial blockade in super obese (BMI ≥ 50 kg/m2), pregnant women, according to the Who classification, whose topographic anatomy is difficult.

DETAILED DESCRIPTION:
Spinal anesthesia is the most commonly used anesthesia method for elective cesarean deliveries. Anesthesiologists may struggle to determine the poorly palpable surface landmarks in super obese (BMI ≥ 50 kg/m2) pregnant women.

The manual palpation technique, preferred in neuraxial anesthesia, may be very difficult in super obese pregnant women due to difficulty identifying bone landmarks. Neuraxial ultrasound examination before spinal anesthesia may help spinal anesthesia performance and decrease the number of attempts in obese parturients.

This study will be a single-center, prospective, randomized, double-blinded trial in a university hospital. Patients scheduled for elective cesarean will be screened for enrollment in the study. The anesthetist administering spinal anesthesia and evaluating the data were blind to the distribution of patient groups. Ultrasonographic examinations were performed by a single investigator trained in this technique who performed more than 60 ultrasound-guided neuraxial blocks.

ELIGIBILITY:
Inclusion Criteria:

* Parturient who will receive selective cesarean delivery under spinal anesthesia
* ASA 3 scheduled for elective sections
* BMI≥50 kg/m2
* Normal singleton pregnancy

  * 37 weeks of gestation

Exclusion Criteria:

* Multiple gestations
* Emergency C-section
* Exist contraindications of spinal anesthesia
* Local anesthetics allergy
* BMI<50 kg/m2
* History of lumbar spinal diseases and lumbar surgery
* Parturient refusal

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — This study only includes pregnant patients who will deliver by elective cesarean section.
Enrollment: 60 (Estimated)
Dates: Start 2024-05-16 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-02 (Estimated)

PRIMARY OUTCOMES:
The success rate of the first puncture | 30 minute
  Success on a single-puncture attempt will be defined as reaching the subarachnoid space on the first insertion of the needle.

SECONDARY OUTCOMES:
Number of skin punctures | 30 minute
  Skin puncture is defined as any separate skin puncture attempt.
Number of needle pass | 30 minute
  Needle pass is defined as skin puncture plus number of redirection attempts
The procedure duration time | 30 minute
  The duration from initiation of location marking by palpation or ultrasound to obtaining free cerebrospinal fluid flow
Time interval to determine needle insertion site | 30 minute
  Time interval between the operator touches the parturient and the completion of the needle insertion point marking
Time taken for spinal injection | 30 minute
  The time interval between the needle insertion to visualization of cerebrospinal spinal fluid in the spinal needle.
Number of puncture levels | 30 minute
  Move to a second lumbar space after 3 needle insertion attempts
Patient satisfaction The procedure duration | 120 minute
  Patients rated their satisfaction as very satisfied, satisfied, or dissatisfied immediately after the procedure.
incidence of complications during puncture | 120 minute
  Incidence of radicular pain, paresthesia, and blood during spinal needle injection
incidence of postoperative headache | 72 hours
  12-72 hours following spinal anesthesia due to CSF leakage
Incidence of hypotension | 2 hours
  A systolic arterial pressure decrease of more than 25% from baseline or less than 90 mmHg
Failure rate of spinal anesthesia | 120 minute
  Number of parturients who need additional analgesic drug or conversion to general anesthesia
dermatome level of sensory block | 10 minute
  thoracic dermatome level of sensory block assessed by pinprick test

CONTACTS AND LOCATIONS:
Overall Officials: Ayşegül Bilge, MD, Principal Investigator — Karaman TRH
Locations (1):
- Karaman Training and Research Hospital, Karaman, Turkey (Türkiye)